CLINICAL TRIAL: NCT01207544
Title: The Effectiveness of Fitball Program Versus Task-oriented Motor Program on Improving Postural Control and Motor Proficiency in Children With Developmental Coordination Disorder
Brief Title: Fitball Program Versus Task-oriented Motor Program on Improving Postural Control in Developmental Coordination Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Collaborators: Kowloon Hospital, Hong Kong (Other)
Responsible Party: Principal Investigator, Marco Yiu-Chung Pang, Associate Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSEARS2009113001
Record Dates: First submitted 2010-09-22; First posted 2010-09-23 (Estimated); Last update posted 2012-11-28 (Estimated); Status verified 2012-11

CONDITIONS: Developmental Coordination Disorder
Keywords: motor; balance; developmental; physiotherapy
MeSH Terms: conditions — Motor Skills Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- fitball program (Experimental): This group will undergo the fitball program consisting of a supervised exercise session once per week for 8 weeks, supplemented by home exercises. The exercise session will be conducted by a qualified physiotherapist.
  Interventions: Behavioral: Fitball exercise
- Task-oriented program (Active Comparator): This group will undergo the task-oriented motor training program consisting of a supervised exercise session once per week for 8 weeks, supplemented by home exercises. The exercise session will be conducted by a qualified physiotherapist.
  Interventions: Behavioral: task-oriented motor training program

INTERVENTIONS:
Behavioral: Fitball exercise — Supervised fitball exercise program session (1 hour per session, 1 session per week, for 8 consecutive weeks), supplemented by daily home exercise program.
  Arms: fitball program
Behavioral: task-oriented motor training program — Task-oriented motor exercise program session (1 hour per session, 1 session per week, for 8 consecutive weeks), supplemented by daily home exercise program.
  Arms: Task-oriented program

SUMMARY:
Children with developmental coordination disorder (DCD) often have poor postural control and motor skills that affect their activities of daily living and participation in school activities. The aim of this randomized controlled trial is to compare the effects of fitball training versus task-oriented motor training for children with DCD.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of DCD according to DSM-IV criteria
* Poor motor skills (Movement Assessment Battery for Children score <15 percentile, or any two or more of subtests in BOT II < 1.5 SD)
* aged between 6-12 years old

Exclusion Criteria:

* have attended treatment for motor problems in the previous 6 months
* any major co-morbid medical / neurological / sensory problems such as moderate to severe mental disability, profound visual or hearing impairment, severe sensory problems, or had any major behavioral problems.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 22 (Actual)
Dates: Start 2010-04; Primary Completion 2011-08 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Brunininks-Oseretsky Test of Motor Proficiency II | Week 0
  Brunininks-Oseretsky Test of Motor Proficiency II is a tool for assessing motor skills.
Brunininks-Oseretsky Test of Motor Proficiency II | Week 8

SECONDARY OUTCOMES:
Sensory Organization Test (SOT) | Week 0
  SOT is a tool for measuring postural stability.
Sensory Organization Test (SOT) | Week 8

CONTACTS AND LOCATIONS:
Overall Officials: Marco YC Pang, PhD, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- The Kowloon Hospital, Kowloon, Hong Kong